CLINICAL TRIAL: NCT01722539
Title: Efficacy and Safety of Sulfadoxine-pyrimethamine or Sulfadoxine-pyrimethamine Plus Piperaquine Regimens Delivered Through Intermittent Preventive Treatment in Schoolchildren of Democratic Republic of Congo: A Randomised Control Trial
Brief Title: Impact IPT With Sulfadoxine-pyrimethamine or Sulfadoxine-pyrimethamine Plus Piperaquine in Schoolchildren
Acronym: PIP-IPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); University of Kinshasa (Other)
Responsible Party: Principal Investigator, Jean-Pierre Van geertruyden, Prof, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PIP-IPT
Record Dates: First submitted 2012-11-03; First posted 2012-11-07 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Healthy
Keywords: intermittent; preventive; treatment; malaria; soil transmitted helminths; schistosomiasis; schoolchildren
MeSH Terms: conditions — Malaria; Schistosomiasis | interventions — fanasil, pyrimethamine drug combination; piperaquine; Albendazole; Praziquantel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sulfadoxine-Pyrimethamine (Experimental): Sulfadoxine-Pyrimethamine every Four months Tablets 500 mg sulfadoxine - 25 mg pyrimethamine will be given as single oral dose of ½ tablets per 10 kg of weigh: 1 tablet for weigh less than 20 kg, 1.5 tablets in 20-29 kg, and 2 tablets for children of weigh 30 or more; Albendazole oral 200 mg will be given to children of 1-2 years and one oral dose of 400 mg to children older than 2 years. The treatment will be repeated at 4-months in the follow-up in accordance with the WHO guideline.
  Praziquantel is a tremacide used for treatment of infections due to schistosomes. Praziquantel will be given as one dose of 40 mg/kg at enrolment and at 12 months follow up.
  Interventions: Drug: Sulfadoxine-pyrimethamine; Drug: Piperaquine; Drug: Albendazole; Drug: Praziquantel
- Sulfadoxine-Pyrimethamine+Piperaquine (Experimental): Sulfadoxine-Pyrimethamine every 4 months Tablets 500 mg sulfadoxine - 25 mg pyrimethamine will be given as single oral dose of ½ tablets per 10 kg of weigh: 1 tablet for weigh less than 20 kg, 1.5 tablets in 20-29 kg, and 2 tablets for children of weigh 30 or more; Piperaquine every four months Piperaquine tablet 320 mg manufactured by Sigma Tau will be used at two treatment doses of 16-24 mg/kg at 24 hours intervals as follows: 1 tablets for weigh 15-19 kg, 1.5 tablets for 20-29 kg, and 2 tablets for 30-39 kg, and 2.5 tablets for 40 kg or more.
  Albendazole oral 200 mg will be given to children of 1-2 years and one oral dose of 400 mg to children older than 2 years. The treatment will be repeated at 4-months in the follow-up in accordance with the WHO guideline.
  Praziquantel is a tremacide used for treatment of infections due to schistosomes. Praziquantel will be given as one dose of 40 mg/kg at enrolment and at 12 months follow up.
  Interventions: Drug: Piperaquine; Drug: Albendazole; Drug: Praziquantel
- Control (Active Comparator): Albendazole oral 200 mg will be given to children of 1-2 years and one oral dose of 400 mg to children older than 2 years. The treatment will be repeated at 4-months in the follow-up in accordance with the WHO guideline.
  Praziquantel is a tremacide used for treatment of infections due to schistosomes. Praziquantel will be given as one dose of 40 mg/kg at enrolment and at 12 months follow up.
  Interventions: Drug: Albendazole; Drug: Praziquantel

INTERVENTIONS:
Drug: Sulfadoxine-pyrimethamine — Tablets 500 mg sulfadoxine - 25 mg pyrimethamine will be given as single oral dose of ½ tablets per 10 kg of weigh: 1 tablet for weigh less than 20 kg, 1.5 tablets in 20-29 kg, and 2 tablets for children of weigh 30 or more
  Other Names: Fansidar
  Arms: Sulfadoxine-Pyrimethamine
Drug: Piperaquine — Piperaquine tablet 320 mg manufactured by Sigma Tau will be used at two treatment doses of 16-24 mg/kg at 24 hours intervals as follows: 1 tablets for weigh 15-19 kg, 1.5 tablets for 20-29 kg, and 2 tablets for 30-39 kg, and 2.5 tablets for 40 kg or more.
  Arms: Sulfadoxine-Pyrimethamine; Sulfadoxine-Pyrimethamine+Piperaquine
Drug: Albendazole — One oral 200 mg will be given to children of 1-2 years and one oral dose of 400 mg to children older than 2 years. The treatment will be repeated at 4-months in the follow-up in accordance with the WHO guideline.
Drug: Praziquantel — Praziquantel is a tremacide used for treatment of infections due to schistosomes. Praziquantel will be given as one dose of 40 mg/kg at enrolment and at 12 months follow up.

SUMMARY:
Considering the facts that: (i) IPT of malaria provides substantial protection against anaemia and malaria in school children (ii); SP resistance has no significant impact on the prophylactic efficacy (iii) SP-PQ is safe and as efficacious as SP: the investigators hypothesize that antimalarial IPT with SP and SP-PQ will improve haemoglobin concentration, reduce anaemia prevalence, malaria incidence and parasitaemia, and improve malnutrition and school performance in school-aged children of Congo.

DETAILED DESCRIPTION:
STUDY RATIONAL The education sector represents a reliable system for malaria control. Intermittent preventive therapy in schoolchildren (IPTsc) is likely the most feasible and appropriate chemoprevention in stable and endemic areas because schoolchildren are usually asymptomatic to malaria infection and are consequently untreated in practice. Therefore, if proven effective, IPTsc would be of direct benefit for the schoolchild, contribute to malaria control at school, and facilitate community-wide the implementation of other control interventions i.e. vector control, Intermittent preventive therapy in infants (IPTi), and prompt diagnosis and treatment (PDT). Nevertheless, evidence about use of IPTsc is not yet substantiated as only two clinical studies have so far been performed on IPTsc in hyper endemic areas. Further clinical trials are warranted in other settings. Through a randomised controlled trial (RCT) we will assess the efficacy and safety, of two IPT regimens versus controls in school children of the DRCongo.

STUDY DRUGS Favourable drugs for use as IPT should balance long half-life against efficacy, safety, tolerability and potentiality for cross-resistance selection.(16) Use of long-acting drugs would result in fewer intake and higher treatment compliance. Sulfadoxine-pyrimethamine is an established used product in the indication of IPT in pregnancy. The drug has further proven safety and tolerability in children in clinical trials. SP is slowly eliminated and allows 60 days antimalaria protection for fully sensitive P. falciparum. Other long-acting drugs available are mefloquine, amodiaquine, and piperaquine. However, due safety concern mefloquine might not be optimal for IPT. Amodiaquine is not suitable for IPT due to its 3 days treatment regimen that may be a concern regarding compliance. Piperaquine has been extensively used for mass prophylaxis and treatment since 1978 in China and other malaria endemic countries of Asia.(20) Piperaquine has a long half-live and points as good IPT candidate in endemic country with SP resistance. For this study sulfadoxine-pyrimethamine combined with piperaquine (SP-PQ) plus will be used. SP and SP-PQ will be given at 4 months intervals in line with the long half-lives (around 20 days) in paediatric patients and for higher treatment compliance,

ELIGIBILITY:
Inclusion Criteria:

* males and females in primary school children,
* anticipated local residence for the study duration,
* signed or thumb-printed informed consent by the parents or guardians and witnessed by an impartial witness (whenever parents/guardians are illiterate)

Exclusion Criteria:

* Children of the 6th primary school year
* Participation in any other investigational drug study (antimalarial or others) during the previous 30 days.
* Known hypersensitivity or serious adverse drug reaction (ADR) to the study drugs.
* Clinical malaria at baseline irrespectively of the severity (World Health Organisation malaria treatment guideline 2010) (Annex III).
* Febrile conditions caused by diseases other than malaria at first visit.
* Clinical symptoms of severe anaemia
* Illness or conditions like hematologic, cardiac, renal, hepatic diseases which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study, including known Glucose 6 phospahate dehydrogenase (G6PD) deficiency and sickle cell (SS form).
* Body weight < 14 kg Children with major chronic infectious diseases (HIV, Tuberculosis, ...)

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 616 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hemoglobin change | Month 0-Month 12
  Change in mean Hb concentration at month 12 of follow-up and anaemia prevalence one year after initial preventive treatment;

SECONDARY OUTCOMES:
Change in mean Hb concentration at month 4 and 8 of follow-up | Month 0 - Month 4 - Month 8
Prevalence of asymptomatic and clinical malaria at baseline & one year after enrolment; | Month 0 Month 12
Prevalence of P. falciparum dihydrofolate reductase (dhfr) and dihydropteroate synthase (dhps) gene mutations at baseline and at month 12 follow-up | Month 0 - Month 12
Clinical (severe) malaria incidence and parasitaemia at month 4, 8, 12; | Month 4, 8 12
Percentages of acute and severe malnourished at month 0, 4, 8, 12 through z-scores, W/H, H/A, and skinfolds | Month 0 - Month 12
Educational achievement, at end of follow-up, and school attendance; | Month 0 - Month 12
Prevalence and risk of environmental and host-related predictors for malaria (re)infections; | Month 0- Month 12
adverse events | Month 0- Months 12

CONTACTS AND LOCATIONS:
Overall Officials: Junior Matangila, MD, Principal Investigator — University of Kinshasa; Pascal Lutumba, MD PhD, Study Director — University of Kinshasa; Joachim Doua, MD, Principal Investigator — Universiteit Antwerpen
Locations (1):
- Mokali health area of Biyela health zone, in Kinshasa province., Kinshasa, Kinshasa Province, Republic of the Congo

REFERENCES:
- [Derived] Doua JY, Matangila J, Lutumba P, Van Geertruyden JP. Intermittent preventive treatment: efficacy and safety of sulfadoxine-pyrimethamine and sulfadoxine-pyrimethamine plus piperaquine regimens in schoolchildren of the Democratic Republic of Congo: a study protocol for a randomized controlled trial. Trials. 2013 Sep 24;14:311. doi: 10.1186/1745-6215-14-311. PMID 24063608